CLINICAL TRIAL: NCT01267058
Title: Single-blind, Clinical Study of the Immunogenicity and Reactogenicity of SB Biologicals' dTpa, pa Vaccines and a Td Vaccine, Given as a Booster Dose to Healthy Adults, From the Age of 18 Years Onwards
Brief Title: Booster Study of Combined Diphtheria-tetanus-acellular Pertussis Vaccine in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 263855/002
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Diphtheria; Pertussis; Tetanus
Keywords: Booster vaccination
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group A (Experimental): Subjects will receive the combined diphtheria, tetanus, acellular pertussis vaccine
  Interventions: Biological: GSK Biologicals' combined diphtheria, tetanus, acellular pertussis vaccine
- Group B (Active Comparator): Subjects will receive the acellular pertussis vaccine and one month later the combined diphtheria and tetanus vaccine
  Interventions: Biological: GSK Biologicals' acellular pertussis vaccine; Biological: Commonwealth Serum Laboratories' combined diphtheria and tetanus vaccine
- Group C (Active Comparator): Subjects will receive the combined diphtheria and tetanus vaccine and one month later the acellular pertussis vaccine
  Interventions: Biological: GSK Biologicals' acellular pertussis vaccine; Biological: Commonwealth Serum Laboratories' combined diphtheria and tetanus vaccine

INTERVENTIONS:
Biological: GSK Biologicals' combined diphtheria, tetanus, acellular pertussis vaccine — Intramuscular, single dose
  Arms: Group A
Biological: GSK Biologicals' acellular pertussis vaccine — Intramuscular, single dose
  Arms: Group B; Group C
Biological: Commonwealth Serum Laboratories' combined diphtheria and tetanus vaccine — Intramuscular, single dose
  Arms: Group B; Group C

SUMMARY:
The aim of the study is to assess the safety and immunogenicity of GlaxoSmithKline Biologicals' (formerly known as SmithKline Beecham Biologicals) combined diphtheria-tetanus-acellular pertussis vaccine in healthy adults, from the age of 18 onwards, in Australia.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of the vaccination
* Written informed consent has been obtained

Exclusion Criteria:

* Evidence of confirmed pertussis disease within the previous 5 years
* History of diphtheria or tetanus vaccination within the past 5 years Females must not be pregnant or lactating They must either surgically sterilized or one year post-menopausal or if they are of childbearing potential, they must be abstinent or have used adequate contraceptive precautions (or one month prior to the booster vaccination, and must agree to continue such precautions for 2 months after completion of the vaccination.
* History of diphtheria or tetanus disease
* History of allergic disease likely to be stimulated by the vaccination
* Major congenital defects or serious chronic illness
* History of progressive neurological disease
* Immunosuppressive therapy
* Any suspected or confirmed immune disorder
* Immunoglobulin therapy or administration of any blood products within the previous three months or during the study period
* Acute febrile illness (>37.5°C, axillary or oral temperature) at the time of planned vaccination
* Administration of an investigational or non registered drug or vaccine within 30 days prior to the start of the present trial
* Simultaneous administration of a vaccine not foreseen by the study protocol, within 30 days prior to the start of the present trial
* Any severe or serious adverse experience having occurred after previous administration of DTP vaccine i.e:

  * an immediate anaphylactic or unacceptable reaction to the investigator's opinion, to a previous dose of diphtheria tetanus pertussis whole-cell vaccine, i.e. :
  * encephalopathy
  * fever > 40.5°C (105°F), rectal temperature, occurring after vaccination with diphtheria tetanus pertussis whole-cell vaccine and not due to another identifiable cause.
  * collapse or shock-like state
  * persistent, inconsolable crying lasting > 3 hours
  * seizures with or without fever
  * systemic allergic or neurologic reactions following a previous dose of tetanus and diphtheria toxoids vaccine
* Exclusion from long term follow-up of antibody persistence : Evidence of confirmed pertussis, diphtheria or tetanus disease or vaccination against these diseases since previous study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 1997-09; Primary Completion 1998-02 (Actual); Study Completion 1998-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and general symptoms | Within the 15-day (Day 0 - Day 14) follow-up period after the first injection

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines | One month after the first injection
Immunogenicity with respect to components of the study vaccines | One month after the second injection
Occurrence of solicited local symptoms and fever | Within the 15-day (Day 0 - Day 14) follow-up period after the second injection
Occurrence of general solicited symptoms to vaccination, other than fever | Within the 15-day (Day 0 - Day 14) follow-up period after each vaccine administration
Occurrence of unsolicited symptoms | Within 31 days (Day 0 - Day 30) after each vaccine administration
Occurrence of serious adverse experiences to vaccination | Within 31 days (Day 0 - Day 30) after each vaccine administration
Immunogenicity with respect to components of the study vaccines | Immediately prior to the booster vaccination
Immunogenicity with respect to components of the study vaccines | One year after the vaccination in a subset of subjects from all the groups
Immunogenicity with respect to components of the study vaccines | 2, 3, 4 and 5 years after the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Cheuvart B, Burgess M, Zepp F, Mertsola J, Wolter J, Schuerman L. Anti-diphtheria antibody seroprotection rates are similar 10 years after vaccination with dTpa or DTPa using a mathematical model. Vaccine. 2004 Dec 2;23(3):336-42. doi: 10.1016/j.vaccine.2004.06.012. PMID 15530678
- [Background] Van Damme P, Burgess M. Immunogenicity of a combined diphtheria-tetanus-acellular pertussis vaccine in adults. Vaccine. 2004 Jan 2;22(3-4):305-8. doi: 10.1016/j.vaccine.2003.08.012. PMID 14670310
- [Background] Turnbull FM, Heath TC, Jalaludin BB, Burgess MA, Ramalho AC. A randomized trial of two acellular pertussis vaccines (dTpa and pa) and a licensed diphtheria-tetanus vaccine (Td) in adults. Vaccine. 2000 Nov 8;19(6):628-36. doi: 10.1016/s0264-410x(00)00252-8. PMID 11090714
- [Result] McIntyre PB, Burgess MA, Egan A, Schuerman L, Hoet B. Booster vaccination of adults with reduced-antigen-content diphtheria, Tetanus and pertussis vaccine: immunogenicity 5 years post-vaccination. Vaccine. 2009 Feb 11;27(7):1062-6. doi: 10.1016/j.vaccine.2008.11.102. Epub 2008 Dec 16. PMID 19095033